CLINICAL TRIAL: NCT00418730
Title: A Phase 2 Multicenter, Randomized, Placebo- and Comparator-Controlled, Double-Blind Parallel Group Study to Evaluate the Safety and Efficacy of Topical NEOSH101 in the Treatment of Androgenetic Alopecia in Men
Brief Title: Efficacy Study of Topical NEOSH101 to Treat Male Pattern Hair Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neosil, Inc. (Industry)
Responsible Party: Andria Langenberg, MD, Vice President, Clinical Development, Neosil, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEOSH101-CLIN-AGA003
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Androgenetic Alopecia
Keywords: androgenetic alopecia; male pattern hair loss; male pattern baldness; androgenetic alopecia or male pattern hair loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: tetrapeptide aldehyde proteasome inhibitor (NEOSH101)
- 2 (Active Comparator)
  Interventions: Drug: tetrapeptide aldehyde proteasome inhibitor (NEOSH101)
- 3 (Placebo Comparator)
  Interventions: Drug: tetrapeptide aldehyde proteasome inhibitor (NEOSH101)

INTERVENTIONS:
Drug: tetrapeptide aldehyde proteasome inhibitor (NEOSH101) — Study preparation (experimental, active comparator, placebo comparator) will be applied twice daily to the scalp for 112 days

SUMMARY:
The purpose of this study is to measure the hair growth response to topical NEOSH101 when applied twice daily to the balding scalp for 16 weeks. One hundred eighty men with Norwood/Hamilton grades III-IV with thinning in the top and center of the scalp will participate. Three equally sized treatment groups (60 men each) will receive either topical NEOSH101 2.0%, minoxidil 5%, or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men, in general good health, aged 18-49 years
* Norwood/Hamilton grades III-IV, with thinning hair in the vertex area

Exclusion Criteria:

* concomitant dermatologic or medical condition(s) which may interfere with the investigator's ability to evaluate the subject's response to the study drug
* treatment with a systemic or locally acting medication which may interfere with the study objectives, such as minoxidil treatment in the 6 months prior to study start, finasteride treatment in the 12 months prior to study start, or treatment with other investigational hair growth products in the 6 months prior to study start

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2007-01; Primary Completion 2007-10 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Hair density, hair growth rate, hair diameter as measured using the TrichoScan method | Through Study Day 197

SECONDARY OUTCOMES:
Assessment score of dermal tolerability | Through Study Day 197
Physician's global assessment score | Through Study Day 197

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Gassmueller, MD, Principal Investigator — Bioskin GmbH
Locations (1):
- bioskin Institute for Dermatological Research and Development GmbH, Hamburg, Germany